CLINICAL TRIAL: NCT02901405
Title: Negative Pressure Dressings Versus Non-negative Pressure Dressing for Wound Care Following Soft Tissue Sarcoma Excision
Brief Title: Negative Pressure Dressing Therapy in Soft Tissue Sarcoma Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was unable to meet recruitment targets
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GN15OR558
Record Dates: First submitted 2016-09-01; First posted 2016-09-15 (Estimated); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Sarcoma; Wound Infection
Keywords: sarcoma; infection; negative pressure
MeSH Terms: conditions — Sarcoma; Wound Infection; Infections | interventions — Negative-Pressure Wound Therapy

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): 120 hours of negative pressure wound therapy (ActiVAC, KCI) applied to a primarily closed ('acute') wound.
  Interventions: Device: Negative Pressure Wound Therapy (ActivVAC, KCI)
- Standard dressings (Active Comparator): Absorbant dressings applied in a standard fashion, i.e. only changed as necessary
  Interventions: Device: Standard dressings

INTERVENTIONS:
Device: Negative Pressure Wound Therapy (ActivVAC, KCI)
  Arms: Negative Pressure Wound Therapy
Device: Standard dressings — Current absorbent dressing is 'tegaderm with absorbent pad' (3M)
  Arms: Standard dressings

SUMMARY:
This randomised controlled trial aims to evaluate the difference in surgical site infection following excision of soft tissue sarcomas. The intervention is a negative wound pressure therapy dressing for 120 hours, the control is standard absorbent dressings

DETAILED DESCRIPTION:
Hypothesis: The application of a negative pressure wound therapy (NPWT) dressing will reduce rates of wound breakdown in patients with resection of soft tissue sarcomas which are primarily closed.

Patients will be randomised into either NPWT or standard absorbent dressings with primary outcome measure of surgical site infection according to the Health Protection Agency guidance. Secondary outcomes are; time to wound dryness, delayed discharge from hospital, adverse events, cost estimation

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing primary soft tissue sarcoma excision which is primarily closed.

Exclusion Criteria:

* Unable to consent
* Children
* Post radiation sarcomas or sarcoma in presence of active infection
* Multiple metastatic disease
* Presence of Endoprosthesis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (proportion) | 30 days
  As diagnosed by independent observer according to the Healthcare Protection Agency (UK) guidelines

SECONDARY OUTCOMES:
Time to wound dryness (nominal scale) | 30 days
  Time to the nearest 12 hour period by which there is no further wound exudate (e.g. staining on dressing)
Delay to discharge form hospital (nominal scale) | 30 days
  Number of additional hospital stays attributable to wound issues
Adverse events (count) | 30 days
  Number of unanticipated events
Cost analysis (comparative nominal scale in £) | 30 days
  Cost analysis to evaluate potential offset of costs for NPWT

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Gupta, MBBS, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom